CLINICAL TRIAL: NCT00364637
Title: Pharmacological Preconditioning Properties of Volatile Anesthetics
Brief Title: Volatile Anesthetics in Cardiac Protection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, DM, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DS/URC/ER/mm 51/DG
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia
Keywords: Sevoflurane; Anesthesia; Troponin; Myocardial Preconditioning; Surgery, Cardiac; Stents; Non-cardiac Surgery; Surgery
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Total intravenous anesthesia (Active Comparator)
  Interventions: Drug: Total intravenous anesthesia
- sevoflurane (Experimental)
  Interventions: Drug: Sevoflurane (Volatile Anesthetic)

INTERVENTIONS:
Drug: Sevoflurane (Volatile Anesthetic)
  Arms: sevoflurane
Drug: Total intravenous anesthesia
  Arms: Total intravenous anesthesia

SUMMARY:
Patients undergoing stenting procedures, or cardiac or non-cardiac surgery could develop myocardial damage as testified by cardiac troponin release.

Sevoflurane (volatile anesthetic), routinely used in cardiac and non-cardiac anesthesia, has cardioprotective properties that could be useful to reduce cardiac damage, as indicated by cardiac troponin release in different contexts:

* stenting procedures (periprocedural administration)
* non-cardiac surgery (during the whole procedure)
* cardiac surgery (during the whole procedure)

DETAILED DESCRIPTION:
Stenting procedures, cardiac and non-cardiac surgical procedures may carry a significant risk of cardiac damage ultimately leading to prolonged hospital stay and even a non-negligible periprocedural mortality rate. According to the American College of Cardiology/American Heart Association Guidelines all anesthetic techniques and drugs have known cardiac effects that should be considered in the perioperative plan. There appears to be no one best myocardium protective anesthetic technique: the choice of anesthesia is best left to the discretion of the anesthesia care team. To date no anesthesiological drug or techniques proved to reduce perioperative morbidity and mortality in cardiac surgery, only Beta-blockers and locoregional analgesia showed improved outcomes after non-cardiac surgery and no study on anesthesiological drugs has been performed in stenting procedures.

Volatile anesthetics, which are commonly used in general anesthesia to induce and maintain hypnosis, analgesia, amnesia and mild muscle relaxation, have been shown to improve post-ischemic recovery at the cellular level, in isolated hearts, and in animals, both through a pharmacological preconditioning and postconditioning action. Whether the cardioprotective effects of volatile anesthetics are clinically applicable and associated with improved cardiac function, ultimately resulting in a better outcome in patients undergoing cardiac surgery, is still debated. No data exist on patients undergoing non-cardiac surgery or stenting procedures.

A recently published meta-analysis including studies considering all volatile anesthetics showed no reduction in myocardial infarction and perioperative death rate. However the newer volatile anesthetics (desflurane and sevoflurane) seem to have more prominent cardioprotective properties and numerous apparently positive reports targeted to surrogate end-points, yet severely underpowered, have appeared in the literature. Of interest, many of these studies were not included in the above cited meta-analysis.

To address the question of whether the choice of an anesthetic regimen might influence patients' outcome we have planned a RCT to determine the impact of sevoflurane on perioperative cardiac damage in patients undergoing cardiac surgery, non-cardiac surgery and stenting procedures.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery
* Non-cardiac surgery
* Stenting procedures

Exclusion Criteria:

* Age < 18 years old
* Not signing written consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Reduce postprocedural cardiac troponin release

SECONDARY OUTCOMES:
Reduce time on mechanical ventilation, Intensive Care Unit (ICU) and hospital stay
mortality

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, MD, Principal Investigator — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia; Alberto Zangrillo, MD, Study Director — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia
Locations (1):
- Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia, Milan, Italy

REFERENCES:
- [Background] Landoni G, Greco T, Biondi-Zoccai G, Nigro Neto C, Febres D, Pintaudi M, Pasin L, Cabrini L, Finco G, Zangrillo A. Anaesthetic drugs and survival: a Bayesian network meta-analysis of randomized trials in cardiac surgery. Br J Anaesth. 2013 Dec;111(6):886-96. doi: 10.1093/bja/aet231. Epub 2013 Jul 12. PMID 23852263
- [Background] Landoni G, Rodseth RN, Santini F, Ponschab M, Ruggeri L, Szekely A, Pasero D, Augoustides JG, Del Sarto PA, Krzych LJ, Corcione A, Slullitel A, Cabrini L, Le Manach Y, Almeida RM, Bignami E, Biondi-Zoccai G, Bove T, Caramelli F, Cariello C, Carpanese A, Clarizia L, Comis M, Conte M, Covello RD, De Santis V, Feltracco P, Giordano G, Pittarello D, Gottin L, Guarracino F, Morelli A, Musu M, Pala G, Pasin L, Pezzoli I, Paternoster G, Remedi R, Roasio A, Zucchetti M, Petrini F, Finco G, Ranieri M, Zangrillo A. Randomized evidence for reduction of perioperative mortality. J Cardiothorac Vasc Anesth. 2012 Oct;26(5):764-72. doi: 10.1053/j.jvca.2012.04.018. Epub 2012 Jun 20. PMID 22726656